CLINICAL TRIAL: NCT03702660
Title: Effect of GIP-receptorantantagonist on Glucagon Plasma Levels After a Meal in Patients With Type 2-diabetes
Brief Title: Effect of GIP After a Meal in Patients With Type 2 Diabetes
Acronym: GA-7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Signe Stensen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GA-7
Record Dates: First submitted 2017-10-30; First posted 2018-10-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — gastric inhibitory polypeptide (3-30)-amide; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GIP(3-30)NH2 (Experimental): GIP receptor antagonist
  Interventions: Other: GIP(3-30)NH2; Other: Peripheral venous cannulation
- Placebo (Placebo Comparator): Placebo (saline infusions)
  Interventions: Other: Peripheral venous cannulation
- GLP-1 (Active Comparator)
  Interventions: Other: Peripheral venous cannulation; Other: GLP-1
- GLP-1 + GIP(3-30)NH2 (Experimental)
  Interventions: Other: GIP(3-30)NH2; Other: Peripheral venous cannulation; Other: GLP-1

INTERVENTIONS:
Other: GIP(3-30)NH2 — Peptide derived from the naturally occuring gut hormone GIP
  Arms: GIP(3-30)NH2; GLP-1 + GIP(3-30)NH2
Other: Peripheral venous cannulation — Intravenous access for infusions
Other: GLP-1 — Peptide infusion
  Arms: GLP-1; GLP-1 + GIP(3-30)NH2

SUMMARY:
The aim of this study is to investigate the effects of antagonising GIP after a meal on plasma levels of glucagon. 10 participants are going through four experimental days each, where they ingest a meal and afterwards receive infusions of either GIP receptor antagonist, GLP-1, GIP receptor antagonist + GLP-1 or placebo (saline) in a randomised order. The primary endpoint of the study is plasma levels of glucagon, which we hypothesize will decrease with infusion of GIP receptor antagonist and/or with infusion of GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians between 18-75 years with diet og Metformin treated type 2-diabetes
* HbA1c < 75 mmol/mol
* BMI > 27 kg/m2
* Stable weight (+/- 5%) during the last 3 months

Exclusion Criteria:

* Treatment with medicine or dietary supplements that cannot the paused for 12 hours
* More than 14 units of alcohol weekly or abuse of drugs
* Liver disease, estimated at plasma ALAT levels > 3 x normal value or INR outside normal range
* Reduced kidney function (estimated at eGFR < 60 ml/min/1,73 m2)
* Severe arteriosclerotic heart disease or heart failure (NYHA III or IV)
* Low red blood cell count (hemoglobin < 8.3 mmol/l
* Special diet or planned weight change during the trial period
* Any disease/condition, which the clinical investigators assess will disturb the participation in the clinical trial

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Glucagon | 8 weeks - 6 months
  Plasma levels of glucagon after a meal in patients with type 2-diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Signe Stensen, MD, Principal Investigator — Center for Diabetes Research
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No